CLINICAL TRIAL: NCT03671564
Title: Phase 1, Open-label, Dose Escalation Study of Milademetan, an Oral MDM2 Inhibitor, to Assess Safety, Tolerability and Pharmacokinetics in Japanese Patients With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Study of Milademetan in Japanese Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS3032-A-J104; 184054 (Registry Identifier: JAPIC CTI)
Record Dates: First submitted 2018-09-04; First posted 2018-09-14 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: Oncology; MDM2; Escalation with overdose control (EWOC)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms | interventions — milademetan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Milademetan (90 mg/Day) (Experimental): Participants who received milademetan 90 mg daily (QD) Day 1 - 14 followed by 14-day rest in a 28-day cycle.
  Interventions: Drug: Milademetan
- Milademetan (120 mg/Day) (Experimental): Participants who received milademetan 120 mg daily (QD) Day 1 - 14 followed by 14-day rest in a 28-day cycle.
  Interventions: Drug: Milademetan
- Milademetan (160 mg/Day) (Experimental): Participants who received milademetan 160 mg daily (QD) Day 1 - 14 followed by 14-day rest in a 28-day cycle.
  Interventions: Drug: Milademetan

INTERVENTIONS:
Drug: Milademetan — Milademetan was administered orally once daily on Days 1 to 14 in a 28-day cycle.
  Other Names: DS-3032b

SUMMARY:
This is a Phase 1, multicenter, open-label study to evaluate safety, tolerability and pharmacokinetics of milademetan in Japanese patients with relapsed or refractory acute myeloid leukemia. The milademetan initial dose will be Level 1: 90 mg. No increase in the milademetan dose will be made in the same participant. Dose-limiting toxicity associated with milademetan occurring at each level will be assessed, and the maximum tolerated dose (MTD) will be decided using a modified continuous reassessment method (mCRM).

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory AML
* AML for which no standard treatment is available
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 2

Exclusion Criteria:

* Acute Promyelocytic Leukemia
* Chronic myelogenous leukemia in blast crisis (BCR-ABL fusion gene positive)
* Presence of central nervous system involvement of leukemia or a history of primary central nervous system leukemia

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (8):
- Japan (8):
  - Japanese Red Cross Narita Hospital, Chiba
  - Kyusyu University Hospital, Fukuoka
  - Gifu Municipal Hospital, Gifu
  - Chugoku Central Hospital, Hiroshima
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Tenri Hospital, Nara
  - NTT Medical Center Tokyo, Tokyo
  - National Hospital Organization Disaster Medical Center, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 14 participants who met all the inclusion criteria and no exclusion criteria were enrolled in study sites in Japan.
Period: Overall Study
Arm/Group | Milademetan (90 mg/Day) | Milademetan (120 mg/Day) | Milademetan (160 mg/Day)
Started | 4 | 6 | 4
Completed | 0 | 0 | 0
Not Completed | 4 | 6 | 4
Not completed — Progressive Disease | 3 | 5 | 3
Not completed — Confirmed TP53 Genotyping Mutation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Demographics and baseline characteristics were assessed in the Enrolled Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Milademetan (90 mg/Day) | Milademetan (120 mg/Day) | Milademetan (160 mg/Day) | Total
Number analyzed (Participants) | 4 | 6 | 4 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 0 | 3
  >=65 years | 3 | 4 | 4 | 11
Age, Continuous [Median (Full Range); unit: years] | 74.5 [57 to 76] | 70.0 [42 to 75] | 71.5 [65 to 75] | 72.0 [42 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 3 | 4
  Male | 4 | 5 | 1 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 6 | 4 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 4 | 6 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) Following Administration of Milademetan in Participants With Relapsed or Refractory Acute Myeloid Leukemia
Description: A dose limiting toxicities (DLTs) is defined as any Grade 3 or higher non-hematological adverse event unless related to the primary disease, course of the primary disease, complications, or concomitant medications, that occurs during the DLT evaluation period (28 days of Cycle 1). The following events will be assessed as DLTs: Grade 4 aspartate aminotransferase (AST)/alanine aminotransferase (ALT), Grade 3 AST/ALT lasting ≥3 days, Grade 3 AST/ALT with Grade ≥2 total bilirubin, and unable to complete at least 75% of the prescribed doses of milademetan in Cycle1 (28 days) as a result of Grade ≥2 events.
Time Frame: First 28 Days of Cycle 1
Population: Dose-limiting toxicities were assessed in the DLT Evaluable Set. 3 participants in the 120-mg cohort were excluded from analysis because study treatment was discontinued before completion of the DLT evaluation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Milademetan (90 mg/Day) | Milademetan (120 mg/Day) | Milademetan (160 mg/Day)
Number analyzed (Participants) | 4 | 3 | 4
Participants | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Following Administration of Milademetan in Participants With Relapsed or Refractory Acute Myeloid Leukemia
Description: Treatment-emergent adverse event (TEAE) is defined as an adverse event that occurs after the first administration, or that worsens relative to the pre-treatment state. An AE is any untoward or unintended sign, symptom, or disease noted in participants who received the study drug, whether it is considered to be related to the study drug or not.
Time Frame: From date of signing of informed consent form up to 30 days after last dose of study drug, up to 1 year
Population: Treatment-emergent adverse events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Milademetan (90 mg/Day) | Milademetan (120 mg/Day) | Milademetan (160 mg/Day)
Number analyzed (Participants) | 4 | 6 | 4
Participants | 4 | 5 | 4

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Milademetan Following Administration of Milademetan in Participants With Relapsed or Refractory Acute Myeloid Leukemia
Description: Maximum Plasma Concentration (Cmax) is defined as the maximum observed plasma concentration and was calculated using non-compartmental analysis.
Time Frame: Days 1 & 14 of Cycle 1: Pre-dose and 1, 2, 3, 6, and 8 hours post-dose (each cycle is 28 days)
Population: Pharmacokinetic parameter was assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Milademetan (90 mg/Day) | Milademetan (120 mg/Day) | Milademetan (160 mg/Day)
Number analyzed (Participants) | 4 | 6 | 4
ng/mL
  Cycle 1, Day 1 | 653 (196) | 1010 (444) | 1380 (540)
  Cycle 1, Day 14: number analyzed (Participants) | 4 | 5 | 4
  Cycle 1, Day 14 | 1090 (327) | 1680 (657) | 2710 (540)

4. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Milademetan Following Administration of Milademetan in Participants With Relapsed or Refractory Acute Myeloid Leukemia
Description: Time of Maximum Plasma Concentration (Tmax) is defined as time of maximum observed plasma concentration and was calculated using non-compartmental analysis.
Time Frame: Days 1 & 14 of Cycle 1: Pre-dose and 1, 2, 3, 6, and 8 hours post-dose (each cycle is 28 days)
Population: Pharmacokinetic parameter was assessed in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | Milademetan (90 mg/Day) | Milademetan (120 mg/Day) | Milademetan (160 mg/Day)
Number analyzed (Participants) | 4 | 6 | 4
hours
  Cycle 1, Day 1 | 4.45 [2.97 to 5.88] | 3.13 [1.92 to 5.92] | 2.54 [2.00 to 8.00]
  Cycle 1, Day 14: number analyzed (Participants) | 4 | 5 | 4
  Cycle 1, Day 14 | 3.02 [2.97 to 3.08] | 2.98 [2.08 to 5.92] | 3.03 [1.87 to 3.17]

5. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) of Milademetan Following Administration of Milademetan in Participants With Relapsed or Refractory Acute Myeloid Leukemia
Description: AUC during 8 hours (AUC8h), AUC during 24 hours (AUC24h), AUC up to the last quantifiable concentration (AUClast), and AUC up to infinity (AUCinf) are presented for Day 1 of Cycle 1 and were assessed using non-compartmental analysis. AUC8h for Day 14 of Cycle 1 is also presented.
Time Frame: Days 1 & 14 of Cycle 1: Pre-dose and 1, 2, 3, 6, and 8 hours post-dose (each cycle is 28 days)
Population: Pharmacokinetic parameter was assessed in the Pharmacokinetic Analysis Set. 2 participants from the Milademetan 90 mg/day and 160 mg/day cohorts for AUC 24 and AUCinf were excluded from the summary as AUC data was not evaluable. 1 participant from Milademetan 120 mg/day cohort for AUC 24 and AUCinf was excluded from the summary as AUC data was not evaluable.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Milademetan (90 mg/Day) | Milademetan (120 mg/Day) | Milademetan (160 mg/Day)
Number analyzed (Participants) | 4 | 6 | 4
ng*h/mL
  Cycle 1 Day 1: AUC8h | 3170 (905) | 4940 (1590) | 6560 (3200)
  Cycle 1 Day 14: AUC8h: number analyzed (Participants) | 4 | 5 | 4
  Cycle 1 Day 14: AUC8h | 6220 (1480) | 10000 (4750) | 15300 (3320)
  Cycle 1 Day 1: AUC24h: number analyzed (Participants) | 2 | 5 | 2
  Cycle 1 Day 1: AUC24h | 8640 (2210) | 12100 (4080) | 15000 (1380)
  Cycle 1 Day 1: AUClast | 8060 (1400) | 11300 (3450) | 14900 (4400)
  Cycle 1 Day 1: AUCinf: number analyzed (Participants) | 2 | 5 | 2
  Cycle 1 Day 1: AUCinf | 13700 (4100) | 18600 (8600) | 22700 (5080)

6. Secondary Outcome: Terminal Elimination Half-Life (T1/2) of Milademetan Following Administration of Milademetan in Participants With Relapsed or Refractory Acute Myeloid Leukemia
Description: Terminal elimination half-life (T1/2) was assessed using non-compartmental analysis.
Time Frame: Day 1 of Cycle 1: Pre-dose and 1, 2, 3, 6, and 8 hours post-dose (each cycle is 28 days)
Population: Pharmacokinetic parameter was assessed in the Pharmacokinetic Analysis Set. 2 participants from the Milademetan 90 mg/day and 160 mg/day cohorts were excluded from the summary as data was not evaluable. 1 participant from Milademetan 120 mg/day cohort was excluded from the summary as data was not evaluable.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Milademetan (90 mg/Day) | Milademetan (120 mg/Day) | Milademetan (160 mg/Day)
Number analyzed (Participants) | 2 | 5 | 2
hours | 15.9 (1.35) | 14.1 (4.27) | 14.6 (4.36)

7. Secondary Outcome: Trough Plasma Concentration (Ctrough) of Milademetan Following Administration of Milademetan in Participants With Relapsed or Refractory Acute Myeloid Leukemia
Description: Trough plasma concentration (Ctrough) was assessed using non-compartmental analysis.
Time Frame: Day 14 of Cycle 1: Pre-dose and 1, 2, 3, 6, and 8 hours post-dose (each cycle is 28 days)
Population: Pharmacokinetic parameter was assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Milademetan (90 mg/Day) | Milademetan (120 mg/Day) | Milademetan (160 mg/Day)
Number analyzed (Participants) | 4 | 5 | 4
ng/mL | 422 (147) | 635 (533) | 769 (221)

8. Secondary Outcome: Number of Participants With Best Response Following Administration of Milademetan in Participants With Relapsed or Refractory Acute Myeloid Leukemia
Description: Best response was defined as the best measured response over all response assessments (complete remission [CR], CR with incomplete hematological recovery [CRi], CR with partial hematological recovery [CRh], partial remission [PR], morphologic leukemia-free state [MLFS], stable disease [SD], or progressive disease [PD]) at all time points after the start of study treatment. The best response will be SD if the response is assessed as SD three or more times consecutively in the protocol-specified evaluation of the antitumor effect. If the response is not assessed as SD three or more times consecutively, the best response will be Not Applicable (unconfirmed SD).
Time Frame: From the start of study treatment to the end of study treatment, up to 1 year
Population: Best Response was assessed on the Efficacy Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Milademetan (90 mg/Day) | Milademetan (120 mg/Day) | Milademetan (160 mg/Day)
Number analyzed (Participants) | 4 | 5 | 3
Participants
  Complete remission (CR) | 0 | 0 | 0
  CR with partial hematological recovery (CRh) | 0 | 0 | 0
  CR with incomplete hematological recovery (CRi) | 0 | 0 | 0
  Partial remission (PR) | 0 | 0 | 0
  Morphologic leukemia-free state (MLFS) | 0 | 1 | 1
  Stable disease (SD) | 1 | 0 | 0
  Progressive disease (PD) | 1 | 1 | 0
  Not applicable (NA) | 2 | 3 | 2
  Not Evaluable (NE) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected from the date of signing the informed consent form up to 30 days after last dose of the study drug, up to 1 year.
Description: An AE is any untoward or unintended sign, symptom, or disease noted in participants who received the study drug, whether it is considered to be related to the study drug or not.
Arm/Group | Milademetan (90 mg/Day) | Milademetan (120 mg/Day) | Milademetan (160 mg/Day)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/4 | 2/6 | 0/4
Other Adverse Events (participants affected / at risk) | 4/4 | 5/6 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Milademetan (90 mg/Day) (N=4) | Milademetan (120 mg/Day) (N=6) | Milademetan (160 mg/Day) (N=4)
Pneumonia (Infections and infestations) | 2 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Milademetan (90 mg/Day) (N=4) | Milademetan (120 mg/Day) (N=6) | Milademetan (160 mg/Day) (N=4)
Pneumonia (Infections and infestations) | 2 | 1 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Skin Infection (Infections and infestations) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 3
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Zinc deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1
Diabetic retinopathy (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1 | 3
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 2 | 1
Oedema peripheral (General disorders) | 1 | 0 | 1
Complication of device insertion (General disorders) | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-07): https://cdn.clinicaltrials.gov/large-docs/64/NCT03671564/Prot_SAP_000.pdf